# Official Title: Feasibility Pilot of Audit and Feedback With Educational Outreach to Align Continuous Pulse Oximetry Use in Stable Bronchiolitis With Evidence and Guideline Recommendations

NCT Number: NCT04178941

Document date: 12/3/2019

#### 1 QUESTIONNAIRE CONSENT LANGUAGE

#### Version 12/03/2019

# 1.1 Text listed in the header of the questionnaire itself

Below you will find a series of questions about the use of continuous pulse oximetry monitoring in bronchiolitis. We are interested in your responses because, in the past few months, you worked on a unit that was part of a study exploring ways to align continuous pulse oximetry use in stable bronchiolitis with national guideline recommendations. In the <a href="attached/linked document">attached/linked document</a>, you will find additional information that may help you decide if you want to take part in the study. Participation is voluntary, and your decision to participate (or not participate) in the research will not affect your performance evaluation or employment. Your response will not be shared with your supervisor.

Completion of the questionnaire below indicates your willingness to participate and serves as your consent.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## 1.2 Detailed text listed on the separate attached/linked document

The Institutional Review Board (IRB) at Children's Hospital of Philadelphia has reviewed this study. The IRB looks at research studies like these and makes sure research subjects' rights and welfare are protected. Below are answers to some questions that you might be wondering about.

### What are the risks of this study?

The main risk of the study is breach of confidentiality, meaning that someone could find out that you completed this questionnaire.

#### Are there any benefits to taking part in this study?

There are no direct benefits. The knowledge gained from this study may help improve the care of children with bronchiolitis.

#### Do you need to give your consent in order to participate?

Yes. Completion of the questionnaire below indicates your willingness to participate and serves as your consent.

#### What happens if you decide not to take part in this study?

Participation in this study is voluntary. You do not have to take part. If you decide not to take part there are no penalties. Your decision to participate (or not participate) in the research will not affect your performance evaluation or employment. Your response will not be shared with your supervisor.

# What about privacy and confidentiality?

We will do our best to keep your personal information private and confidential. However, we cannot guarantee absolute confidentiality. Your personal information may be disclosed if required by law. People from oversight agencies and organizations such as the Department of Health and Human Services and the Office for Human Research Protections may also look at your study records. The results of this study may be shown at meetings and published in journals to inform other health professionals. We will keep your identity private in any publication or presentation. By law, we are

required to protect your private information. The investigators and staff involved in the study will keep your private information collected for the study strictly confidential.

A Certificate of Confidentiality (CoC) issued by the NIH covers this research. A CoC helps protect your identifiable information and biological samples. A CoC protects your private information from all legal proceedings. Unless you consent, information from this research study that identifies you will not be shared outside this research. Specifically, (1) no one can be forced to share your identifiable information for a lawsuit, and (2) your information can't be used as evidence even if there is a court subpoena. The CoC does not prevent some disclosures. The researchers can't refuse requests for information from those funding this research. The National Institutes of Health may need information to assess this project. You can still share information about yourself. You can also freely discuss your involvement in this research. The researchers must disclose things required by law. This includes suspected child abuse and neglect, harm to self or others, or communicable diseases.

# Who is funding this research study?

Children's Hospital of Philadelphia and The National Institutes of Health are funding this study.

#### What if you have other questions about the study?

If you have questions about this study or how your data will be used, email the study doctor, Dr. Bonafide at <a href="mailto:bonafide@email.chop.edu">bonafide@email.chop.edu</a> or call his office at 267-426-2901. If you have questions about your rights or if you have a complaint, you can call the Children's Hospital of Philadelphia IRB Office at 215-590-2830.